CLINICAL TRIAL: NCT04971863
Title: In-vivo Behavior of Asqelio Monofocal Biaspheric Intraocular Lens. Two-year Follow-up
Brief Title: In-vivo Behavior of Asqelio Monofocal Biaspheric Intraocular Lens
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: ASQM012021
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-02

CONDITIONS: Cataract; Intraocular Lens Complication
Keywords: posterior capsule opacitication; incidence
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clareon Monofocal IOL: Patients bilaterally implanted with the Clareon monofocal IOL
- Asqelio Monofocal IOL: Patients bilaterally implanted with the Asqelio monofocal IOL

SUMMARY:
This is a study to evaluate the 24 month postoperative incidence and intensity of posterior capsular opacity in patients submitted to cataract surgery and implanted with a hydrophobic monofocal IOL.

DETAILED DESCRIPTION:
This study is a two-arm masked clinical evaluation study of incidence of PCO after successful bilateral cataract surgery with implantation of a monofocal IOL. Subjects will be assessed 24 months after IOL implantation. Clinical evaluations will include incidence of adverse events, patient satisfaction questionnaire, as well as measurements of visual performance, optical quality, presence and intensity of PCO, presence and intensity of IOL glistening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 22 years or older submitted to cataract surgery in at least 1 eye and implanted with Asqelio monofocal or Clareon monofocal IOL

Exclusion Criteria:

* Any pathology reducing potential best-corrected visual acuity beyond 0.30 LogMAR, including amblyopia, severe corneal dystrophy, diabetic retinopathy, extremely shallow anterior chamber, microphthalmos, retinal detachment, severe recurrent anterior or posterior segment inflammation of unknown ethiology, iris neovascularization, uncontrolled glaucoma, clinically significant macular degeneration, or pseudoexfoliation diagnosis.
* Previous ocular surgery
* Rubella
* Surgery motivated by traumatic cataract
* Ocular trauma or refractive surgery
* Any other systemic or ocular condition that, in the investigator's opinion, should exclude the subject from study
* Requiring additional procedures due to intraoperatory complications, mechanical or surgical interventions for manipulating the pupil, excessive iris movility, significant vitreous loss, significant, anterior chamber hyphema, capsular annular breakage, or any other unrecognized ocular conditions that might compromise IOL positioning, as well as impossibility of locate the IOL in the capsular bag due to surgical complications.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects submitted to non-traumatic cataract surgery in at least 1 eye at the Hospital La Fé of Valencia, Spain
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Posterior capsular opacity | 24 months after IOL implantation
  Incidence of PCO
Intensity of Posterior capsular opacity | 24 months after IOL implantation
  Intensity of PCO determined using LOCSIII Classification System

SECONDARY OUTCOMES:
Visual acuity | 1 month, 6 months, 12 months and 24 months after IOL implantation
  Best corrected distance visual acuity in LogMAR units using the ETDRS chart
Refraction | 1 month, 6 months, 12 months and 24 months after IOL implantation
  Residual refractive error in diopters determined objectively
Optical quality | 24 months after IOL implantation
  Higher-order wavefront aberrations determined using a clinical wavefront analyzer
Incidence of Glistening | 24 months after IOL implantation
  Incidence of IOL glistening
Intensity of Glistening | 24 months after IOL implantation
  Intensity of IOL glistening

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico la Fe, Valencia, Spain

REFERENCES:
- [Derived] Hervas-Ontiveros A, Espana-Gregori E, Fresno-Canada C, Butron-Ruiz R, Cervino A. Posterior Capsular Opacification and Glistening in Hydrophobic Monofocal Biaspheric Intraocular Lens Two Years After Implantation: A Case Control Study. J Ophthalmol. 2024 Dec 31;2024:3520219. doi: 10.1155/joph/3520219. eCollection 2024. PMID 39781444